CLINICAL TRIAL: NCT02002910
Title: Japan Study of Distal Evaluation of Functional Significance of Intra-arterial Stenosis Narrowing Effect
Status: Completed | Type: Observational
Sponsor: Associations for Establishment of Evidence in Interventions (Other)
Responsible Party: Sponsor
Other Study IDs: J-DEFINE
Record Dates: First submitted 2013-10-28; First posted 2013-12-06 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
Keywords: iFR; FFR; Medical Economy; physiological assessment; SYNTAX score
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate whether instantaneous wave-Free Ratio(iFR)/Fractional Flow Reserve(FFR) guided treatment strategy makes the postulated treatment strategy by Coronary Angiogram(CAG) guide change and to analyze the cost-effectiveness of its dual diagnosis.

To investigate difference between SYNTAX score evaluated CAG and functional SYNTAX score evaluated physiological assessment of coronary stenosis and its clinical effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age>=20 years old.
* Patient who can understand informed consent of the clinical study and signed the consent.
* Patient who is adaptable to CAG and/or coronary revascularization
* Patient who has evaluated stenotic lesion (stenosis>50% in visual judgment) by CAG at main epicardial vessel and its branch or who suspected to have it.

Exclusion Criteria:

* Patient with known contraindications to Adenosine Triphosphate(ATP) and/or papaverine hydrochloride
* Target vessel diameter<=2.0mm
* Lesion with Chronic Total Occlusion(CTO) (registration allowed if other branch has stenosis more than 50% in visual judgment)
* Patient with temporary/permanent artificial pacemaker implantation, left bundle branch block, second-degree and third-degree atrioventricular block.
* Acute Myocardial Infarction(AMI) patient
* Patient who is disqualified for FFR and coronary revascularization by the investigator.
* Lesion is disqualified for Percutaneous Coronary Intervention(PCI) by the investigator.
* Patient who has critical valvular disease of heart. (moderate or severe Aortic valve stenosis(AS)/Aortic Regurgitation(AR)/Mitral Stenosis(MS)/Mitral Regurgitation(MR)）
* Patient with a prior Coronary Artery Bypass Graft(CABG) on target vessel.
* Patient with severe renal dysfunction. (serum creatinine>=2.0mg/dl)
* Patient on hemodialysis.
* Body weight>=200kg
* Patient who needs ventricular assist device to ensure hemodynamic stability (heart rate<50/min, SBP<90mmHg)
* Patient who expects to live less than 2 years at the registration
* Patient with contraindications to an antithrombotic therapy or an anticoagulant therapy.
* Patient who is poor compliance with drug treatment.
* Patient who is allergic to contrast agent.
* Left Ventricular Ejection Fraction(LVEF)>=30%
* Patient who has the history of PCI with Drug-Eluting Stent(DES) in recent 3 months before registration.
* Patient who has the history of PCI with Bare Metal Stent(BMS) or Plain Old Balloon Atherectomy(POBA) in recent 1 year before registration.
* Patient who has possibility of pregnancy, under breast-feeding and positive pregnancy test in 14days prior to the PCI.
* Patients with inadequacy to join this clinical study.
* Patient who has been enrolled any other clinical study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who is adaptable to CAG and/or coronary revascularization
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Medical economy | 1 year after the procedure
  To evaluate the healthcare cost-effectiveness in QALY（Quality Adjusted Life Year）converted by Japanese functional score ; Quality of Life(QOL) questionnaire (EQ-5D) and the cost postulated by CAG strategy with its iFR/FFR hybrid strategy.
  To collect the healthcare cost related MACCE at the timing of 6 and 12 months FU point. (Included emergency visit) To collect QOL questionnaire (EQ-5D) at the timing of just after the treatment and 12 months follow up point.
Physiological assessment | baseline pocedure
  Alteration in treatment protocol. Change in SYNTAX score.

SECONDARY OUTCOMES:
Incidence of major adverse cardiac and cerebrovascular events(MACCE) | 1year after the pocedure
  MACCE include all-cause death, cerebrovascular accident(CVA), myocardial infarction(MI), and repeat revascularization.
correlated analysis | baseline pocedure
  Area under receiver-operating characteristic curve(ROC) Classification agreement between iFR and FFR in this registry, Demonstrated using the area under the receiver-operating characteristic curve(FFR cut-off 0.8 or 0.75).
evaluation of variance | beseline procedure
  Treatment categorization disagreements of iFR and FFR are analyzed by multi-variable analysis processing to calculate Characteristic factors.

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, M.D, Study Chair
Locations (1):
- NPO Associations for Establishment of Evidence in Interventions, Minato, Tokyo, Japan